CLINICAL TRIAL: NCT00258726
Title: Immunogenicity and Safety of Live Attenuated Varicella Vaccine in 12 and 18 Month-old Children, With and Without Concomitant Administration of Measles-Mumps-Rubella Vaccine
Brief Title: Immune Responses to Two Dose Varivax +/- MMR-II
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-073
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-04

CONDITIONS: Measles; Mumps; Rubella; Varicella
Keywords: Measels, Mumps, Varicella, Rubella, vaccine, children
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — Chickenpox Vaccine

INTERVENTIONS:
Biological: MMR-II
Biological: Pro-Quad
Biological: Varivax

SUMMARY:
This study will test the safety and how well the body's immune system responds to a live, but weakened varicella (chickenpox) vaccine, known as Varivax, given with and without ProQuad, another measles, mumps, rubella, and varicella virus vaccine (MMR-II). One hundred five healthy children will be enrolled in the study when they are 12 months old. All subjects will be vaccinated at 12 months of age and some subjects will receive a second vaccination at 18 months of age. All subjects will participate for 1 year. This study is a single-site, two-year trial with post-licensure vaccines.

DETAILED DESCRIPTION:
This clinical trial is a phase I/II exploratory immunogenicity and safety study of live attenuated Varicella (Varivax), Measles-Mumps-Rubella (MMR-II), or combination Varicella/Measles, Mumps/Rubella (Pro-Quad) vaccines administered to healthy children at 12 and 18 months of age. A total of 105 healthy children, 12 months old at the time of study entry, will be recruited from the Palo Alto Medical Foundation clinics in Palo Alto, Fremont and Los Altos, California. The study is designed to focus on time of primary Varivax immunization and immunologic benefits of a two-dose vaccine regimen compared to a single Varivax dose. In addition, the investigators will evaluate the use of Varivax with and without concomitant administration of the MMR-II, further measuring immunologic responses to a two-dose MMR-II regimen. The first study objective is to determine the immunogenicity of one dose of Varivax administered at 12 versus 18 months of age. Participants will receive either MMR vaccine and Varivax, or ProQuad depending on availability of the vaccines. Immunogenicity to be measured as humoral responses utilizing plaque reduction neutralization (PRN) assay for measles and gpELISA for varicella antibodies, and T cell immunity determined by flow cytometric T cell assays. The second study objective is to determine the immunogenicity of administering two doses of Varivax and MMR-II to children at 12 and 18 months of age compared with children receiving one dose of MMR-II at 12 months and one dose of Varivax at 12 or 18 months of age. Participants will receive either MMR vaccine and Varivax, or ProQuad depending on availability of the vaccines. The third study objective is to determine the safety of administering two doses of Varivax and MMR-II to children at 12 and 18 months of age. Participants will receive either MMR vaccine and Varivax, or ProQuad depending on availability of the vaccine. Study personnel with documentation of all adverse events and serious adverse events will monitor safety using parental memory aids and telephone follow-up. The investigators hypothesize that infants receiving Varivax or ProQuad at 12 months of age will have comparable humoral immune responses to infants receiving the vaccine at 18 months of age, but that T cell immunity will be higher in those vaccinated at 18 months of age. In addition, infants receiving 2 doses of Varivax or ProQuad will have higher humoral and cell mediated immune responses compared with children receiving only one dose of Varivax or ProQuad. This hypothesis would explain the post-licensure observations that breakthrough disease is higher in those vaccinated at 12 versus 15 months of age and in children who received one vaccination compared with two. The investigators predict that there will be no differences in the humoral immune responses when measles is given concomitantly with Varivax compared to Varivax alone, but the immunosuppressive effects of the measles virus can influence effects on T cell immunity. It is expected that two doses of Varivax or Proquad will be well tolerated and that there will be fewer systemic adverse reactions after the second dose. The Varivax package insert reports that the incidence of injection site redness and swelling was slightly higher post dose 2, but the incidence of systemic clinical complaints was lower post dose 2. The incidence of adverse experiences both locally and systemically following a second dose of ProQuad was equal to or less than those reactions seen after the first dose. The investigators will evaluate the incidence of injection site reactogenicity to confirm these findings.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants 12 months (+ 4 weeks) of age.
2. Free of obvious health problems as established by medical history and clinical examination before entering into the study. This includes all chronic health problems and immunodeficiencies.
3. Parent/legal guardian has provided signed, written informed consent.
4. Parent/legal guardian expected to be available for entire study.
5. Parent/legal guardian can be reached by telephone.

Exclusion Criteria:

1. Former premature infants (<36 weeks).
2. Birth weight < 2500 grams.
3. Significant underlying chronic illness.
4. Immunodeficiency disease or use of immunosuppressive therapy by the participant.
5. Any other condition that in the clinical judgment of the investigator might interfere with vaccine evaluation.
6. Allergy to any components of the vaccine, including anaphylaxis or anaphylaxoid reaction to neomycin or eggs for MMR-II, and/or hypersensitivity to gelatin and anaphylaxis or anaphylaxoid reaction to neomycin for Varivax.
7. Plans for participation in another clinical trial with an investigational drug or vaccine for the duration of this study.
8. Blood products within 3 months prior to initial enrollment.
9. Previous receipt of MMR and Varivax or ProQuad.

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States